CLINICAL TRIAL: NCT00647101
Title: Open Multicenter Study on the Efficacy of Xalatan at 3 Months as First-line Therapy in Naive Patients With Ocular Hypertension (OH) or Open Angle Glaucoma (OAG), Based on Initial Intraocular Pressure (IOP): 20 mmHg Less Than or Equal to IOP Less Than 24 mmHg, IOP Greater Than or Equal to 24 mmHg
Brief Title: A Study to Assess the Efficacy of 3 Months of Latanoprost Treatment in Reducing the Intraocular Pressure in Patients With Ocular Hypertension or Open-angle Glaucoma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6111002; X-FIL
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2008-03

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Latanoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Latanoprost group (Experimental)
  Interventions: Drug: Latanoprost

INTERVENTIONS:
Drug: Latanoprost — Latanoprost 0.005% drops: 1 drop in the diseased eye(s) in the evening for 3 months

SUMMARY:
The purpose of this study is to evaluate the effect of latanoprost on intraocular pressure reduction in patients with ocular hypertension or open-angle glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* A patient with an IOP greater than or equal to 20 mmHg related to unilateral or bilateral OH or OAG (primary open angle glaucoma, pseudo-exfoliative glaucoma, and pigmentary glaucoma), after a visual field exam
* Naive patients (i.e. never having been treated) and requiring treatment initiation

Exclusion Criteria:

* A patient with OH or OAG currently on treatment
* A patient with OH or OAG previously treated (regardless of the date treatment was discontinued)
* A patient with traumatic, inflammatory, or neovascular glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2003-12; Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Change in IOP after 3 months of treatment in absolute values (mmHg) compared to baseline IOP | 3 months

SECONDARY OUTCOMES:
Change in IOP after 3 months of treatment in relative values (percentage of decrease) compared to baseline IOP | 3 months
Proportion of patients after 3 months of treatment with a relative reduction in IOP of greater than or equal to 30%, and greater than or equal to 10% | 3 months
Change in IOP after 1 month of treatment in absolute (mmHg) and relative values (percentage of decrease) relative to baseline IOP | 1 month
Proportion of patients after 1 month of treatment with a relative reduction in IOP of greater than or equal to 30%, and greater than or equal to 10% | 1 month
Proportion of patients after 3 months of treatment achieving the following target IOP values: IOP less than or equal to 21 mmHg, IOP less than or equal to 18 mmHg, IOP less than or equal to 15 mmHg | 3 months
Proportion of patients after 1 month of treatment achieving the following target IOP values: IOP less than or equal to 21 mmHg, IOP less than or equal to 18 mmHg, IOP less than or equal to 15 mmHg | 1 month
Occurrence of adverse events on latanoprost, local tolerability analysis by clinical exam | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (149):
- France (149):
  - Pfizer Investigational Site, Albi
  - Pfizer Investigational Site, Ambert
  - Pfizer Investigational Site, Amboise
  - Pfizer Investigational Site, Angers
  - Pfizer Investigational Site, Antibes
  - Pfizer Investigational Site, Aubenas
  - Pfizer Investigational Site, Belfort
  - Pfizer Investigational Site, Bergerac
  - Pfizer Investigational Site, Bernay
  - Pfizer Investigational Site, Béthune
  - Pfizer Investigational Site, Béziers
  - Pfizer Investigational Site, Blagnac
  - Pfizer Investigational Site, Bordeaux
  - Pfizer Investigational Site, Bougival
  - Pfizer Investigational Site, Boulogne-Billancourt
  - Pfizer Investigational Site, Brest
  - Pfizer Investigational Site, Bry-sur-Marne
  - Pfizer Investigational Site, Carentan
  - Pfizer Investigational Site, Cenon
  - Pfizer Investigational Site, Chamalières
  - Pfizer Investigational Site, Chantilly
  - Pfizer Investigational Site, Chartres
  - Pfizer Investigational Site, Châteaubriant
  - Pfizer Investigational Site, Châteaulin
  - Pfizer Investigational Site, Clermont-Ferrand
  - Pfizer Investigational Site, Condom
  - Pfizer Investigational Site, Coulommiers
  - Pfizer Investigational Site, Courbevoie
  - Pfizer Investigational Site, Creil
  - Pfizer Investigational Site, Deauville
  - Pfizer Investigational Site, Deuil-la-Barre
  - Pfizer Investigational Site, Douai
  - Pfizer Investigational Site, Draveil
  - Pfizer Investigational Site, Enghien-les-Bains
  - Pfizer Investigational Site, Épernay
  - Pfizer Investigational Site, Fontaine
  - Pfizer Investigational Site, Fréjus
  - Pfizer Investigational Site, Gennevilliers
  - Pfizer Investigational Site, Gradignan
  - Pfizer Investigational Site, Grasse
  - Pfizer Investigational Site, Grenoble
  - Pfizer Investigational Site, Guingamp
  - Pfizer Investigational Site, Haguenau
  - Pfizer Investigational Site, Herblay-sur-Seine
  - Pfizer Investigational Site, Hyères
  - Pfizer Investigational Site, Issy-les-Moulineaux
  - Pfizer Investigational Site, Ivry-sur-Seine
  - Pfizer Investigational Site, Jarville-la-Malgrange
  - Pfizer Investigational Site, Joigny
  - Pfizer Investigational Site, Juvisy-sur-Orge
  - Pfizer Investigational Site, La Rochelle
  - Pfizer Investigational Site, La Talaudière
  - Pfizer Investigational Site, La Trinité
  - Pfizer Investigational Site, Landerneau
  - Pfizer Investigational Site, Langon
  - Pfizer Investigational Site, Lannion
  - Pfizer Investigational Site, Laon
  - Pfizer Investigational Site, Le Creuzot
  - Pfizer Investigational Site, Le Havre
  - Pfizer Investigational Site, Le Mans
  - Pfizer Investigational Site, Le Peage de Rousillon
  - Pfizer Investigational Site, Le Quesnoy
  - Pfizer Investigational Site, Lesneven
  - Pfizer Investigational Site, Lille
  - Pfizer Investigational Site, Livry-Gargan
  - Pfizer Investigational Site, Lunel
  - Pfizer Investigational Site, Lunéville
  - Pfizer Investigational Site, Luxeuil-les-Bains
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Maisons-Laffitte
  - Pfizer Investigational Site, Marcq-en-Barœul
  - Pfizer Investigational Site, Marignanne
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Meyzieu
  - Pfizer Investigational Site, Montauban
  - Pfizer Investigational Site, Montceau-les-Mines
  - Pfizer Investigational Site, Montpellier
  - Pfizer Investigational Site, Mulhouse
  - Pfizer Investigational Site, Nantes
  - Pfizer Investigational Site, Nice
  - Pfizer Investigational Site, Niort
  - Pfizer Investigational Site, Nîmes
  - Pfizer Investigational Site, Nogent-sur-Marne
  - Pfizer Investigational Site, Noyon
  - Pfizer Investigational Site, Orléans
  - Pfizer Investigational Site, Oullins
  - Pfizer Investigational Site, Pantin
  - Pfizer Investigational Site, Paray-le-Monial
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Pau
  - Pfizer Investigational Site, Pauillac
  - Pfizer Investigational Site, Perros Girec
  - Pfizer Investigational Site, Périgueux
  - Pfizer Investigational Site, Pézenas
  - Pfizer Investigational Site, Poissy
  - Pfizer Investigational Site, Poitiers
  - Pfizer Investigational Site, Pont-de-Chéruy
  - Pfizer Investigational Site, Pornic
  - Pfizer Investigational Site, Port-de-Bouc
  - Pfizer Investigational Site, Quimper
  - Pfizer Investigational Site, Reims
  - Pfizer Investigational Site, Rochefort
  - Pfizer Investigational Site, Romilly-sur-Seine
  - Pfizer Investigational Site, Saint Savine
  - Pfizer Investigational Site, Saint-Brieuc
  - Pfizer Investigational Site, Saint-Chamond
  - Pfizer Investigational Site, Saint-Dié
  - Pfizer Investigational Site, Saint-Etienne
  - Pfizer Investigational Site, Saint-Gaudens
  - Pfizer Investigational Site, Saint-Lô
  - Pfizer Investigational Site, Saint-Michel-sur-Orge
  - Pfizer Investigational Site, Saintes
  - Pfizer Investigational Site, Salon-de-Provence
  - Pfizer Investigational Site, Sartrouville
  - Pfizer Investigational Site, Sens
  - Pfizer Investigational Site, Sessiney Pariset
  - Pfizer Investigational Site, Sète
  - Pfizer Investigational Site, Soissons
  - Pfizer Investigational Site, Strasbourg
  - Pfizer Investigational Site, Suresnes
  - Pfizer Investigational Site, Talence
  - Pfizer Investigational Site, Thiers
  - Pfizer Investigational Site, Toulon
  - Pfizer Investigational Site, Toulouse
  - Pfizer Investigational Site, Tourcoing
  - Pfizer Investigational Site, Tournefeuille
  - Pfizer Investigational Site, Tours
  - Pfizer Investigational Site, Tremblay-en-France
  - Pfizer Investigational Site, Trélissac
  - Pfizer Investigational Site, Triel-sur-Seine
  - Pfizer Investigational Site, Troyes
  - Pfizer Investigational Site, Valenciennes
  - Pfizer Investigational Site, Vannes
  - Pfizer Investigational Site, Vauvert
  - Pfizer Investigational Site, Veauche
  - Pfizer Investigational Site, Velaux
  - Pfizer Investigational Site, Vendargues
  - Pfizer Investigational Site, Vénissieux
  - Pfizer Investigational Site, Viarmes
  - Pfizer Investigational Site, Vienne
  - Pfizer Investigational Site, Villeneuve-d'Ascq
  - Pfizer Investigational Site, Villeneuve-la-Garenne
  - Pfizer Investigational Site, Villeneuve-Saint-Georges
  - Pfizer Investigational Site, Villeparisis
  - Pfizer Investigational Site, Villepinte
  - Pfizer Investigational Site, Villiers-le-Bel
  - Pfizer Investigational Site, Vizille
  - Pfizer Investigational Site, Voiron
  - Pfizer Investigational Site, Wattrelos

REFERENCES:
- [Derived] Denis P, Baudouin C, Bron A, Nordmann JP, Renard JP, Rouland JF, Sellem E, Amrane M. First-line latanoprost therapy in ocular hypertension or open-angle glaucoma patients: a 3-month efficacy analysis stratified by initial intraocular pressure. BMC Ophthalmol. 2010 Feb 24;10:4. doi: 10.1186/1471-2415-10-4. PMID 20181282
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6111002&StudyName=A%20Study%20to%20Assess%20the%20Efficacy%20of%203%20Months%20of%20Latanoprost%20Treatment%20in%20Reducing%20the%20Intraocular%20Pressure%20in%20Patients%20with%20Ocular%20Hyp